CLINICAL TRIAL: NCT05513794
Title: Prospective Data Collect Study for Development of Neurimelanin Image Analysis System
Brief Title: Prospective Study for Neuromelanin Image Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heuron Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: qMT-PD-02
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2024-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient group (Experimental): Patient with parkinson disease
  Interventions: Device: MRI Imaging
- Healthy volunteer group (Experimental): Healthy volunteer
  Interventions: Device: MRI Imaging

INTERVENTIONS:
Device: MRI Imaging — Neuromelanin sequence imaging

SUMMARY:
In order to develop an image analysis system that automatically detects and quantifies neuromelanin, this study aims to construct a database of a wide sample by collecting brain MRI neuromelanin images prospectively.

ELIGIBILITY:
Parkinsin group

Inclusion Criteria:

* Adults over 19 years old
* Those who have clinically shown Parkinson's symptoms such as tremor, Rigidity, Bradykinesa and gait disturbance and are scheduled to take MRI scans
* Dopamine transporter imaging shows a significant decrease in visual dopamine intake
* A person who can read and understand the description and informed consent form
* Upon hearing and fully understanding the detailed explanation of this clinical trial, a person who has voluntarily decided to participate and agreed in writing to comply with the precautions

Exclusion Criteria:

* Patient with a history of claustrophobia and mental illness;
* Patient with metallic substances in the body
* Any female subject who is likely to be pregnant who does not agree to contraception in a medically permitted manner during this clinical trial period
* Pregnant or lactating women
* Other cases where the investigator judged that it is difficult to participate in the study;

Healthy volunteer group

Inclusion Criteria:

* Adults over 19 years old
* A person who has no family history or diagnostic history of movement disorders;
* A person with a score of 8 or higher on the CCSIT(cross cultural smell identification test)
* A person with a score of 27 or higher on the MMSE Test
* No Parkinson's symptoms on a neurological examination
* Upon hearing and fully understanding the detailed explanation of this clinical trial, a person who has voluntarily decided to participate and agreed in writing to comply with the precautions

Exclusion Criteria:

* Patient with a history of central nervous system disease or cognitive disorder
* Patient with a history of claustrophobia and mental illness;
* Patient with metallic substances in the body
* Any female subject who is likely to be pregnant who does not agree to contraception in a medically permitted manner during this clinical trial period
* Pregnant or lactating women
* Other cases where the investigator judged that it is difficult to participate in the study;

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-07-02 (Actual)

PRIMARY OUTCOMES:
Differences in Neuromelanin Volume by Age | Within 1 weeks after enrollment
  Descriptive Statistics for Neuromelanin Volume Measured by MRI Image by Age

SECONDARY OUTCOMES:
Differences in Neuromelanin Volume by group | Within 1 weeks after enrollment
  Descriptive Statistics for Neuromelanin Volume Measured by MRI Image by group

CONTACTS AND LOCATIONS:
Overall Officials: Phil Hyu Lee, M.D.pH.D, Principal Investigator — Severance Hospital, Yonsei University Health System
Locations (3):
- South Korea (3):
  - Inje University Sanggye Paik Hospital, Seoul, nowon-gu
  - Severance Hospital, Yonsei University Health System, Seoul, Seodaemun gu
  - Yong-in Severance Hospital, Yonsei University Health System, Gyeonggi-do, yongin-si

IPD SHARING:
Plan to Share IPD: No